CLINICAL TRIAL: NCT06176677
Title: Comparative Evaluation of Training Effectiveness Between Commercial Videolaryngoscope and Low-Cost Self Built Laryngoscope With Hyperangulated Blade
Brief Title: Use of a Low-cost Video Laryngoscope on Manikin
Status: Completed | Type: Observational
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Responsible Party: Principal Investigator, Alessandro Tani, Principal investigator, Azienda USL Toscana Nord Ovest
Other Study IDs: AVNO2024-1
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Airway Management

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Videolaryngoscope — We set as endpoint the time from insertion of each laryngoscope through the mouth to complete visualization of the glottis (T1) and the time to complete intubation manoeuvre(T2)
Device: Boroscope — We set as endpoint the time from insertion of each laryngoscope through the mouth to complete visualization of the glottis (T1) and the time to complete intubation manoeuvre(T2)

SUMMARY:
Videolaryngoscopy has become essential in airway management, providing improved glottis visualization and reducing intubation attempts. Proficiency in using videolaryngoscopes, especially those with hyperangulated blades, is crucial for challenging intubation cases. However, successful intubation with hyperangulated blades requires continuous training due to their unique shape. Despite the benefits, the high cost of commercial videolaryngoscopes limits their use, prompting the exploration of a cost-effective alternative-a self-built laryngoscope using a USB borescope. The study aims to compare its training effectiveness with a commercial hyperangulated blade videolaryngoscope, emphasizing accessible training options. The evaluation involves testing both devices on a Laerdal® intubation mannequin, focusing on the time to glottis visualization and the time to complete intubation.

DETAILED DESCRIPTION:
Videolaryngoscopy has become integral in airway management, providing improved visualization of the glottis and reducing the number of intubation attempts. Proficiency in the use of videolaryngoscopes is essential, particularly in cases of difficult intubation. Videolaryngoscopes equipped with hyperangulated blades facilitate enhanced visualization, even in the most challenging scenarios. However, successful intubation using these blades requires adequate training due to their unique shape. While hyperangulated blades offer excellent views around the curvature of the tongue, their upward perspective from the base of the tongue can pose challenges in tube delivery. Therefore, continuous training is essential to achieve proficiency with these particular blades.

Despite the advantages, the high cost of commercially available videolaryngoscopes poses a barrier to regular use and training, especially in resource-limited settings. This study introduces a cost-effective alternative-a self-built laryngoscope using a Universal Serial Bus (USB) borescope. The objective is to compare its training effectiveness with that of a commercial hyperangulated blade videolaryngoscope, underscoring the significance of accessible training options.

The Glidescope videolaryngoscope and a custom-built laryngoscope equipped with a USB borescope blade will undergo testing. The evaluation will be conducted by 30 emergency and operating room personnel following a brief training course in videolaryngoscopy, using a Laerdal® intubation mannequin. Both devices will utilize size 4 hyperangulated blades with identical curvature angles. Assessment endpoints will encompass the duration required for glottis visualization and the time needed for the entire intubation process.

ELIGIBILITY:
Inclusion Criteria: emergency and operating room personnel who have participated and completed the videolaryngoscopy course -

Exclusion Criteria: any temporary or permanent physical impediment to performing the requested maneuver or not having participated or completed the videolaryngoscopy course

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 doctors and nurses in the emergency area and operating room
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
compare the effectiveness of training between a commercial videolaryngoscope and a low cost videolaryngoscope | one hour
  Compare the training effectiveness between a commercial videolaryngoscope and a low-cost videolaryngoscope by measuring the time from the insertion of each laryngoscope through the mouth to the complete visualization of the glottis (T1) and the time taken for the entire intubation maneuver (T2) in the manikin, among 30 emergency and operating room operators .

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Tani, MD, Principal Investigator — area Vasta Toscana Nordovest
Locations (1):
- Santa Maria Maddalena Hospital, Volterra, Pisa, Italy

REFERENCES:
- [Background] Tani A, Vagheggini G, Tudisco S, Del Colombo V, Mannelli E, Lehle J. Use of low-cost modified laryngoscope for training in videolaryngoscopy. A comparison between a Macintosh modified laryngoscope and Stortz C MAC 8403XDK: a manikin study. Minerva Anestesiol. 2022 Jan-Feb;88(1-2):85-86. doi: 10.23736/S0375-9393.21.15998-X. Epub 2021 Sep 16. No abstract available. PMID 34527409